CLINICAL TRIAL: NCT07312123
Title: Effect of Oral Alpha-Lipoic Acid, Vitamin E, and Vitamin B Combination on Symptoms and Function in Carpal Tunnel Syndrome Following Carpal Tunnel Surgery
Brief Title: A Study to See Whether Taking a Mix of Vitamins Can Help Adults Recover Better After Surgery for Carpal Tunnel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universiti Sains Malaysia (Other)
Collaborators: BREGO Life Sciences Sdn Bhd (Unknown)
Responsible Party: Principal Investigator, NURHAKIM BIN IBRAHIM, medical officer, master student in orthopedic, Hospital Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/25060535; NMRR ID-25-01261-KS3 (Other: National Medical Research Register by National Institutes of Health , Ministry of Health Malaysia)
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; median nerve compression; vitamin e; peripheral nerve entrapment
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Thioctic Acid; Vitamin E; Vitamin B Complex

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Antioxidant Supplement Group (Experimental)
  Interventions: Dietary Supplement: Alpha-Lipoic Acid, Vitamin E, and Vitamin B Complex
- Control Group (Active Comparator)
  Interventions: Dietary Supplement: combination vitamin b1,b6 b12

INTERVENTIONS:
Dietary Supplement: Alpha-Lipoic Acid, Vitamin E, and Vitamin B Complex — An oral dietary supplement containing a combination of alpha-lipoic acid, Vitamin E, and Vitamin B complex administered once daily for the study duration. The supplement is provided in capsule form and is intended to support nerve health through antioxidant and neuroprotective effects in patients with Carpal Tunnel Syndrome.
  Arms: Oral Antioxidant Supplement Group
Dietary Supplement: combination vitamin b1,b6 b12 — An oral Vitamin B complex supplement administered once daily for the study duration. This intervention serves as the active comparator for conservative treatment of Carpal Tunnel Syndrome.
  Arms: Control Group

SUMMARY:
Carpal Tunnel Syndrome (CTS) is a common condition that causes numbness, tingling, pain, and weakness in the hand due to compression of the median nerve at the wrist. It can affect daily activities, work performance, and quality of life. While surgery is effective in severe cases, many patients with mild to moderate CTS are initially treated with non-surgical options such as splinting and medications. However, the effectiveness of oral supplements for CTS remains uncertain.

This clinical study aims to evaluate whether an oral combination of alpha-lipoic acid, Vitamin E, and Vitamin B complex can safely reduce symptoms and improve hand function in patients with Carpal Tunnel Syndrome. These supplements are believed to have antioxidant, anti-inflammatory, and nerve-protective properties, which may help reduce nerve irritation and improve nerve recovery.

Participants in this study will be randomly assigned to receive either the oral supplement combination or a comparator treatment. The study is single-blinded, meaning participants will not know which treatment they are receiving. Symptoms such as pain, numbness, and hand function will be assessed over a defined follow-up period using clinical evaluation and standardized questionnaires.

The main hypothesis of this study is that patients receiving the oral combination of alpha-lipoic acid, Vitamin E, and Vitamin B will experience greater improvement in symptoms and functional outcomes compared to those who do not receive the combination, without significant side effects.

The results of this study may help determine whether this oral supplement combination can be used as an effective and safe conservative treatment option for patients with Carpal Tunnel Syndrome, potentially reducing the need for invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* Subjects with symptoms and physical examination of CTS
* Patients with CTS going for CT release

Exclusion Criteria:

* Pregnant or breast-feeding women
* Patients with history of trauma in the dominant hand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-12-08 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) score | baseline to 12 and 24 weeks

SECONDARY OUTCOMES:
Change in Pain Intensity Measured by Visual Analog Scale | baseline to 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: nurhakim bin ibrahim, Principal Investigator — Hospital Pakar Universiti Sains Malaysia
Locations (1):
- Hospital Pakar Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia